CLINICAL TRIAL: NCT01529346
Title: A Randomized, Double-blind, Double-dummy, Parallel Group, Placebo Controlled Study Assessing The Efficacy Of Single Doses Of Pf-05089771 For The Treatment Of Postoperative Dental Pain Using Ibuprofen 400 Mg As Positive Control
Brief Title: Efficacy Of PF-05089771 In Treating Postoperative Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3291009
Record Dates: First submitted 2011-12-13; First posted 2012-02-08 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Dental Pain
Keywords: Postoperative dental pain
MeSH Terms: interventions — PF-05089771; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- PF-05089771 1600 mg (Experimental)
  Interventions: Drug: PF-05089771; Other: Placebo
- PF-05089771 450 mg (Experimental)
  Interventions: Drug: PF-05089771; Other: Placebo
- PF-05089771 150 mg (Experimental)
  Interventions: Drug: PF-05089771; Other: Placebo
- Ibuprofen 400 mg (Active Comparator)
  Interventions: Drug: Ibuprofen; Other: Placebo
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-05089771 — A single dose of PF-05089771 1600 mg oral solution administered once to the subject on Day 1 postoperatively
  Arms: PF-05089771 1600 mg
Other: Placebo — Placebo tablets for ibuprofen: 2 X 200 mg placebo tablets administered orally once to the subject on Day 1 postoperatively
  Arms: PF-05089771 1600 mg
Drug: PF-05089771 — A single dose of PF-05089771 450 mg oral solution administered once to the subject on Day 1 postoperatively
  Arms: PF-05089771 450 mg
Other: Placebo — Placebo tablets for ibuprofen: 2 X 200 mg placebo tablets administered orally once to the subject on Day 1 postoperatively
  Arms: PF-05089771 450 mg
Drug: PF-05089771 — A single dose of PF-05089771 150 mg oral solution administered once to the subject on Day 1 postoperatively
  Arms: PF-05089771 150 mg
Other: Placebo — Placebo tablets for ibuprofen: 2 X 200 mg placebo tablets administered orally once to the subject on Day 1 postoperatively
  Arms: PF-05089771 150 mg
Drug: Ibuprofen — 2 X 200 mg tablets of ibuprofen administered orally once to the subject on Day 1 postoperatively
  Arms: Ibuprofen 400 mg
Other: Placebo — Placebo solution for PF-05089771: A single dose of Placebo solution administered once to the subject on Day 1 postoperatively
  Arms: Ibuprofen 400 mg
Other: Placebo — Placebo solution for PF-05089771:A single dose of Placebo solution administered once to the subject on Day 1 postoperatively
  Arms: Placebo
Other: Placebo — Placebo tablets for Ibuprofen: 2 X 200 mg placebo tablets administered orally once to the subject on Day 1 postoperatively
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the overall pain relief of a single dose of PF-05089771 against placebo following third molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Oral surgery having removed 2 unilateral third molar teeth.
* Pre-dose pain intensity score (100 mm VAS [VAS]) of at least 50mm within 5 hours of oral surgery
* Pre-dose pain intensity score of moderate or severe within 5 hours of oral surgery

Exclusion Criteria:

* Presence or known history of any clinically significant hematological, hepatic, renal, endocrine, cardiovascular, neurological, psychiatric, gastrointestinal, pulmonary, allergic (including known drug hypersensitivities or allergies, but excluding untreated asymptomatic seasonal allergy) or any metabolic disorder that may increase risk associated with study participation, investigational drug administration or may interfere with interpretation of study results.
* Prior use of any type of analgesic or NSAID within 5-half lives of that drug or less before taking the first dose of study medication, except for anesthesia for the procedure.
* Active dental infection at the time of surgery.
* Recent (within the previous 12 months) history of chronic analgesic or tranquiliser dependency.
* Any significant oral surgery complication at the time of surgery or in the immediate postoperative period, or oral surgery that has lasted more than 30 minutes (time from first incision to last suture placement).

Subjects who smoke more than 1 pack (20 cigarettes) per day, more than 3 cigars per day or use smokeless tobacco on a daily basis are excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 235 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2012-06-25 (Actual); Study Completion 2012-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Central Texas Oral Surgery Associates, Austin, Texas
  - Premier Research Group Limited, Austin, Texas
  - PPD Development, LP, Austin, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291009&StudyName=Efficacy%20Of%20PF-05089771%20In%20Treating%20Postoperative%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-05089771 150 mg: Single oral dose of PF-05089771 150 milligram (mg) -dispersion along with 2 placebo tablets matched to ibuprofen 200 mg tablet orally following unilateral surgical extraction of two-third molars, one of which was a partial or full bony mandibular impaction. Study treatment was administered within 5 hours post-surgery when the pain intensity reached the required moderate to severe level (score of 2 or greater on a 4-point categorical pain severity rating scale and a score of at least 50 millimeter [mm] on a 100 mm Visual Analog Scale [VAS] pain severity rating scale).
- PF-05089771 450 mg: Single oral dose of PF-05089771 450 mg -dispersion along with 2 placebo tablets matched to ibuprofen 200 mg tablet orally following unilateral surgical extraction of two-third molars, one of which was a partial or full bony mandibular impaction. Study treatment was administered within 5 hours post-surgery when the pain intensity reached the required moderate to severe level (score of 2 or greater on a 4-point categorical pain severity rating scale and a score of at least 50 mm on a 100 mm VAS pain severity rating scale).
- PF-05089771 1600 mg: Single oral dose of PF-05089771 1600 mg -dispersion along with 2 placebo tablets matched to ibuprofen 200 mg tablet orally following unilateral surgical extraction of two-third molars, one of which was a partial or full bony mandibular impaction. Study treatment was administered within 5 hours post-surgery when the pain intensity reached the required moderate to severe level (score of 2 or greater on a 4-point categorical pain severity rating scale and a score of at least 50 mm on a 100 mm VAS pain severity rating scale).
- Ibuprofen: Single oral dose of 2 ibuprofen 200 mg tablets (equivalent to ibuprofen 400 mg) along with placebo matched to PF-05089771-dispersion orally following unilateral surgical extraction of two-third molars, one of which was a partial or full bony mandibular impaction. Study treatment was administered within 5 hours post-surgery when the pain intensity reached the required moderate to severe level (score of 2 or greater on a 4-point categorical pain severity rating scale and a score of at least 50 mm on a 100 mm VAS pain severity rating scale).
- Placebo: Single oral dose of 2 placebo tablets matched to ibuprofen tablets along with placebo matched to PF-05089771-dispersion orally following unilateral surgical extraction of two-third molars, one of which was a partial or full bony mandibular impaction. Study treatment was administered within 5 hours post-surgery when the pain intensity reached the required moderate to severe level (score of 2 or greater on a 4-point categorical pain severity rating scale and a score of at least 50 mm on a 100 mm VAS pain severity rating scale).
Period: Overall Study
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Started | 55 | 54 | 54 | 36 | 36
Completed | 53 | 53 | 52 | 36 | 36
Not Completed | 2 | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo | Total
Number analyzed (Participants) | 55 | 54 | 54 | 36 | 36 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (6.1) | 23.3 (4.9) | 24.0 (4.9) | 22.7 (4.7) | 24.2 (6.4) | 23.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 15 | 9 | 13 | 69
  Male | 41 | 36 | 39 | 27 | 23 | 166

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Relief From 0 to 6 Hours (TOTPAR[6])
Description: TOTPAR(6) was defined as the total area under pain relief (PR) curve through first 6 hours after dosing, calculated using trapezoidal rule. PR was assumed to be 0 at 0 hour. PR assessed on a 5-point categorical scale: 0(none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete), at different time points during study up to 6 hours. Total score range for TOTPAR(6): 0 (worst) to 24 (best), higher value indicated greater degree of PR. Posterior mean, standard deviation were estimated based on analysis of covariance (ANCOVA) model with non-informative priors within outlier robust Bayesian framework.
Time Frame: 0 to 6 hours
Population: Full Analysis Set (FAS): all randomized participants who received at least (>=) 1 dose of study treatment and had >=1 evaluable (more than or equal to [>=] 90 minutes post-dose) PR score. Participants who received rescue medication prior to 90 minutes were not included in FAS. Missing data were imputed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
units on a scale | 6.94 (0.898) | 6.21 (0.915) | 7.00 (0.906) | 14.43 (1.110) | 4.37 (1.082)

2. Secondary Outcome: Number of Participants With Peak Pain Relief (PPR)
Description: PPR was defined as the highest PR score achieved at any time point during the evaluation period, prior to rescue medication. PR was assessed on a 5-point categorical scale: 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete).
Time Frame: 0 to 24 hours
Population: FAS included all randomized participants who received >=1 dose of study treatment and had >=1 evaluable (>=90 minutes post-dose) pain relief score. Participants who received rescue medication prior to 90 minutes were not included in FAS.
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
participants
  None | 13 | 13 | 15 | 1 | 9
  A Little | 11 | 11 | 6 | 4 | 10
  Some | 10 | 10 | 11 | 1 | 9
  A Lot | 4 | 9 | 6 | 11 | 4
  Complete | 16 | 11 | 15 | 19 | 4

3. Secondary Outcome: Pain Relief (PR) Score
Description: PR was assessed on a 5-point categorical scale; 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete).
Time Frame: 15, 30, 45, 60, 90 minutes, 2, 3, 4, 6, 8, 24 hours
Population: FAS included all randomized participants who received >=1 dose of study treatment and had >=1 evaluable (>=90 minutes post-dose) pain relief score. Analysis excluded influential outliers. Participants who received rescue medication prior to 90 minutes were not included in FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
units on a scale
  15 Minutes | 0.55 (0.11) | 0.72 (0.11) | 0.65 (0.11) | 0.54 (0.14) | 0.63 (0.14)
  30 Minutes | 0.77 (0.15) | 1.09 (0.14) | 0.86 (0.15) | 1.36 (0.18) | 0.70 (0.18)
  45 Minutes | 0.90 (0.15) | 1.26 (0.15) | 0.98 (0.15) | 1.89 (0.18) | 0.87 (0.18)
  60 Minutes | 0.99 (0.16) | 1.13 (0.16) | 1.10 (0.16) | 2.09 (0.19) | 0.79 (0.19)
  90 Minutes | 1.12 (0.16) | 1.06 (0.16) | 1.11 (0.16) | 2.42 (0.20) | 0.73 (0.20)
  2 Hours | 1.19 (0.19) | 1.23 (0.19) | 1.14 (0.19) | 2.48 (0.22) | 0.70 (0.23)
  3 Hours | 1.57 (0.18) | 1.63 (0.19) | 1.61 (0.18) | 2.85 (0.20) | 0.98 (0.26)
  4 Hours | 1.95 (0.18) | 1.79 (0.20) | 1.89 (0.18) | 3.07 (0.19) | 1.46 (0.28)
  6 Hours | 2.02 (0.21) | 1.92 (0.24) | 2.18 (0.21) | 2.97 (0.21) | 2.07 (0.36)
  8 Hours | 2.21 (0.24) | 2.20 (0.28) | 2.08 (0.22) | 2.65 (0.22) | 2.38 (0.39)
  24 Hours | 3.59 (0.16) | 3.20 (0.18) | 3.40 (0.14) | 3.15 (0.17) | 2.96 (0.24)
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; 15 Minutes: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; Least Squares (LS) Mean Difference = -0.08, 90% CI 2-sided [-0.38 to 0.22], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.09, 90% CI 2-sided [-0.20 to 0.39], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.02, 90% CI 2-sided [-0.28 to 0.32], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.09, 90% CI 2-sided [-0.41 to 0.24], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: PF-05089771 150 mg vs Placebo; 30 Minutes: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.06, 90% CI 2-sided [-0.32 to 0.44], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.39, 90% CI 2-sided [0.01 to 0.77], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.16, 90% CI 2-sided [-0.22 to 0.54], Standard Error of Mean 0.23
Statistical Analysis 8: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.66, 90% CI 2-sided [0.24 to 1.07], Standard Error of Mean 0.25
Statistical Analysis 9: Comparison: PF-05089771 150 mg vs Placebo; 45 Minutes: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.02, 90% CI 2-sided [-0.37 to 0.42], Standard Error of Mean 0.24
Statistical Analysis 10: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 0.39, 90% CI 2-sided [-0.00 to 0.78], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 0.11, 90% CI 2-sided [-0.29 to 0.50], Standard Error of Mean 0.24
Statistical Analysis 12: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 1.02, 90% CI 2-sided [0.59 to 1.45], Standard Error of Mean 0.26
Statistical Analysis 13: Comparison: PF-05089771 150 mg vs Placebo; 60 Minutes: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.20, 90% CI 2-sided [-0.21 to 0.62], Standard Error of Mean 0.25
Statistical Analysis 14: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 0.34, 90% CI 2-sided [-0.07 to 0.76], Standard Error of Mean 0.25
Statistical Analysis 15: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 0.30, 90% CI 2-sided [-0.11 to 0.72], Standard Error of Mean 0.25
Statistical Analysis 16: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 1.30, 90% CI 2-sided [0.85 to 1.75], Standard Error of Mean 0.27
Statistical Analysis 17: Comparison: PF-05089771 150 mg vs Placebo; 90 Minutes: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.39, 90% CI 2-sided [-0.04 to 0.81], Standard Error of Mean 0.26
Statistical Analysis 18: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 0.32, 90% CI 2-sided [-0.10 to 0.75], Standard Error of Mean 0.26
Statistical Analysis 19: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 0.38, 90% CI 2-sided [-0.05 to 0.81], Standard Error of Mean 0.26
Statistical Analysis 20: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 1.69, 90% CI 2-sided [1.22 to 2.15], Standard Error of Mean 0.28
Statistical Analysis 21: Comparison: PF-05089771 150 mg vs Placebo; 2 Hours: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.50, 90% CI 2-sided [0.01 to 0.99], Standard Error of Mean 0.30
Statistical Analysis 22: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 0.54, 90% CI 2-sided [0.05 to 1.03], Standard Error of Mean 0.30
Statistical Analysis 23: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 0.45, 90% CI 2-sided [-0.04 to 0.94], Standard Error of Mean 0.30
Statistical Analysis 24: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 1.79, 90% CI 2-sided [1.26 to 2.31], Standard Error of Mean 0.32
Statistical Analysis 25: Comparison: PF-05089771 150 mg vs Placebo; 3 Hours: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.59, 90% CI 2-sided [0.06 to 1.11], Standard Error of Mean 0.32
Statistical Analysis 26: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 0.64, 90% CI 2-sided [0.11 to 1.17], Standard Error of Mean 0.32
Statistical Analysis 27: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 0.63, 90% CI 2-sided [0.11 to 1.15], Standard Error of Mean 0.32
Statistical Analysis 28: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 1.87, 90% CI 2-sided [1.33 to 2.40], Standard Error of Mean 0.32
Statistical Analysis 29: Comparison: PF-05089771 150 mg vs Placebo; 4 Hours: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.49, 90% CI 2-sided [-0.07 to 1.05], Standard Error of Mean 0.34
Statistical Analysis 30: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 0.33, 90% CI 2-sided [-0.24 to 0.91], Standard Error of Mean 0.35
Statistical Analysis 31: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 0.43, 90% CI 2-sided [-0.13 to 0.98], Standard Error of Mean 0.34
Statistical Analysis 32: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 1.61, 90% CI 2-sided [1.05 to 2.17], Standard Error of Mean 0.34
Statistical Analysis 33: Comparison: PF-05089771 150 mg vs Placebo; 6 Hours: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = -0.05, 90% CI 2-sided [-0.74 to 0.64], Standard Error of Mean 0.42
Statistical Analysis 34: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = -0.15, 90% CI 2-sided [-0.86 to 0.56], Standard Error of Mean 0.43
Statistical Analysis 35: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = 0.11, 90% CI 2-sided [-0.57 to 0.80], Standard Error of Mean 0.42
Statistical Analysis 36: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = 0.90, 90% CI 2-sided [0.22 to 1.58], Standard Error of Mean 0.41
Statistical Analysis 37: Comparison: PF-05089771 150 mg vs Placebo; 8 Hours: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = -0.17, 90% CI 2-sided [-0.93 to 0.59], Standard Error of Mean 0.46
Statistical Analysis 38: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = -0.18, 90% CI 2-sided [-0.98 to 0.62], Standard Error of Mean 0.48
Statistical Analysis 39: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = -0.30, 90% CI 2-sided [-1.05 to 0.45], Standard Error of Mean 0.45
Statistical Analysis 40: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = 0.27, 90% CI 2-sided [-0.47 to 1.02], Standard Error of Mean 0.45
Statistical Analysis 41: Comparison: PF-05089771 150 mg vs Placebo; 24 Hours: repeated measures model included baseline pain intensity, treatment, time, the treatment by time interaction and the time by baseline pain intensity interaction as fixed effects. The unstructured covariance matrix was used to estimate the variances and covariance within participant across time points; Test type: Superiority or Other; LS Mean Difference = 0.63, 90% CI 2-sided [0.15 to 1.11], Standard Error of Mean 0.29
Statistical Analysis 42: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.24, 90% CI 2-sided [-0.27 to 0.74], Standard Error of Mean 0.30
Statistical Analysis 43: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.44, 90% CI 2-sided [-0.03 to 0.91], Standard Error of Mean 0.28
Statistical Analysis 44: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.19, 90% CI 2-sided [-0.30 to 0.67], Standard Error of Mean 0.29

4. Secondary Outcome: Pain Intensity Difference (PID)
Description: PID was calculated as pain intensity at baseline (baseline pain severity score range 2 [moderate] to 3 [severe]) minus pain intensity at the respective post-baseline visit (pain severity score range 0 [none] to 3 [severe]). Total possible score range for PID: -1 (worst) to 3 (best).
Time Frame: 15, 30, 45, 60, 90 minutes, 2, 3, 4, 6, 8, 24 hours
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
units on a scale
  15 Minutes | 0.12 (0.06) | 0.34 (0.06) | 0.21 (0.07) | 0.16 (0.08) | 0.14 (0.08)
  30 Minutes | 0.32 (0.10) | 0.57 (0.10) | 0.42 (0.10) | 0.72 (0.12) | 0.13 (0.12)
  45 Minutes | 0.34 (0.11) | 0.62 (0.11) | 0.44 (0.11) | 0.93 (0.13) | 0.22 (0.13)
  60 Minutes | 0.38 (0.11) | 0.47 (0.11) | 0.41 (0.11) | 1.01 (0.14) | 0.28 (0.14)
  90 Minutes | 0.38 (0.12) | 0.36 (0.12) | 0.45 (0.12) | 1.32 (0.15) | 0.06 (0.15)
  2 Hours | 0.45 (0.14) | 0.38 (0.14) | 0.46 (0.14) | 1.35 (0.16) | 0.05 (0.17)
  3 Hours | 0.74 (0.13) | 0.76 (0.14) | 0.82 (0.13) | 1.56 (0.14) | 0.18 (0.20)
  4 Hours | 1.02 (0.14) | 0.92 (0.15) | 1.03 (0.14) | 1.69 (0.14) | 0.52 (0.22)
  6 Hours | 1.05 (0.15) | 0.96 (0.17) | 1.09 (0.15) | 1.65 (0.14) | 0.82 (0.26)
  8 Hours | 1.08 (0.18) | 1.11 (0.21) | 1.01 (0.17) | 1.40 (0.16) | 0.76 (0.29)
  24 Hours | 2.15 (0.12) | 1.73 (0.15) | 2.00 (0.11) | 1.76 (0.13) | 1.70 (0.19)
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = -0.02, 90% CI 2-sided [-0.19 to 0.14], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.20, 90% CI 2-sided [0.03 to 0.37], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.07, 90% CI 2-sided [-0.10 to 0.24], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 0.02, 90% CI 2-sided [-0.16 to 0.21], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.20, 90% CI 2-sided [-0.06 to 0.45], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.44, 90% CI 2-sided [0.19 to 0.70], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.29, 90% CI 2-sided [0.04 to 0.54], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 0.59, 90% CI 2-sided [0.32 to 0.87], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 0.12, 90% CI 2-sided [-0.16 to 0.40], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 0.40, 90% CI 2-sided [0.12 to 0.68], Standard Error of Mean 0.17
Statistical Analysis 11: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 0.23, 90% CI 2-sided [-0.05 to 0.50], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; LS Mean Difference = 0.71, 90% CI 2-sided [0.40 to 1.01], Standard Error of Mean 0.18
Statistical Analysis 13: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 0.10, 90% CI 2-sided [-0.19 to 0.40], Standard Error of Mean 0.18
Statistical Analysis 14: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 0.19, 90% CI 2-sided [-0.10 to 0.49], Standard Error of Mean 0.18
Statistical Analysis 15: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 0.13, 90% CI 2-sided [-0.16 to 0.43], Standard Error of Mean 0.18
Statistical Analysis 16: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; LS Mean Difference = 0.74, 90% CI 2-sided [0.41 to 1.06], Standard Error of Mean 0.20
Statistical Analysis 17: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 0.33, 90% CI 2-sided [0.01 to 0.64], Standard Error of Mean 0.19
Statistical Analysis 18: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 0.31, 90% CI 2-sided [-0.01 to 0.62], Standard Error of Mean 0.19
Statistical Analysis 19: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 0.39, 90% CI 2-sided [0.08 to 0.71], Standard Error of Mean 0.19
Statistical Analysis 20: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; LS Mean Difference = 1.26, 90% CI 2-sided [0.92 to 1.61], Standard Error of Mean 0.21
Statistical Analysis 21: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 0.40, 90% CI 2-sided [0.04 to 0.76], Standard Error of Mean 0.22
Statistical Analysis 22: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 0.33, 90% CI 2-sided [-0.03 to 0.69], Standard Error of Mean 0.22
Statistical Analysis 23: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 0.41, 90% CI 2-sided [0.05 to 0.77], Standard Error of Mean 0.22
Statistical Analysis 24: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; LS Mean Difference = 1.30, 90% CI 2-sided [0.92 to 1.68], Standard Error of Mean 0.23
Statistical Analysis 25: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 0.55, 90% CI 2-sided [0.16 to 0.95], Standard Error of Mean 0.24
Statistical Analysis 26: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 0.57, 90% CI 2-sided [0.17 to 0.97], Standard Error of Mean 0.24
Statistical Analysis 27: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 0.63, 90% CI 2-sided [0.24 to 1.03], Standard Error of Mean 0.24
Statistical Analysis 28: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; LS Mean Difference = 1.38, 90% CI 2-sided [0.97 to 1.78], Standard Error of Mean 0.24
Statistical Analysis 29: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 0.50, 90% CI 2-sided [0.08 to 0.92], Standard Error of Mean 0.25
Statistical Analysis 30: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 0.41, 90% CI 2-sided [-0.03 to 0.84], Standard Error of Mean 0.26
Statistical Analysis 31: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 0.51, 90% CI 2-sided [0.09 to 0.93], Standard Error of Mean 0.25
Statistical Analysis 32: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; LS Mean Difference = 1.17, 90% CI 2-sided [0.75 to 1.59], Standard Error of Mean 0.25
Statistical Analysis 33: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = 0.23, 90% CI 2-sided [-0.27 to 0.72], Standard Error of Mean 0.30
Statistical Analysis 34: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = 0.14, 90% CI 2-sided [-0.37 to 0.65], Standard Error of Mean 0.31
Statistical Analysis 35: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = 0.27, 90% CI 2-sided [-0.23 to 0.77], Standard Error of Mean 0.30
Statistical Analysis 36: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; LS Mean Difference = 0.82, 90% CI 2-sided [0.33 to 1.31], Standard Error of Mean 0.30
Statistical Analysis 37: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = 0.32, 90% CI 2-sided [-0.24 to 0.89], Standard Error of Mean 0.34
Statistical Analysis 38: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = 0.34, 90% CI 2-sided [-0.25 to 0.94], Standard Error of Mean 0.36
Statistical Analysis 39: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = 0.25, 90% CI 2-sided [-0.31 to 0.80], Standard Error of Mean 0.34
Statistical Analysis 40: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; LS Mean Difference = 0.64, 90% CI 2-sided [0.08 to 1.19], Standard Error of Mean 0.33
Statistical Analysis 41: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.45, 90% CI 2-sided [0.07 to 0.83], Standard Error of Mean 0.23
Statistical Analysis 42: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.04, 90% CI 2-sided [-0.36 to 0.44], Standard Error of Mean 0.24
Statistical Analysis 43: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.31, 90% CI 2-sided [-0.07 to 0.68], Standard Error of Mean 0.22
Statistical Analysis 44: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; LS Mean Difference = 0.06, 90% CI 2-sided [-0.32 to 0.45], Standard Error of Mean 0.23

5. Secondary Outcome: Summed Pain Intensity Difference (SPID)
Description: SPID: area under the PID effect curve from 0 to 6 hours (SPID[6]) and 0 to 24 hours (SPID[24]). AUC was calculated using the trapezoidal rule. Total score range: -6 (worst) to 18 (best) for SPID(6), and -24 (worst) to 72 (best) for SPID(24). Higher value of SPID indicated greater degree of pain relief. PID was calculated as pain intensity at baseline minus pain intensity at the respective post-baseline visit. Pain intensity was assessed on a categorical scale ranging from 0 (none), 1 (mild), 2 (moderate) and 3 (severe).
Time Frame: 0 to 6 hours; 0 to 24 hours
Population: FAS included all randomized participants who received >=1 dose of study treatment and had >=1 evaluable (>=90 minutes post-dose) pain relief score. Analysis excluded influential outliers. Participants who received rescue medication prior to 90 minutes were not included in FAS. Missing data were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
units on a scale
  SIPD(6) | 2.52 (0.63) | 2.14 (0.63) | 2.79 (0.64) | 7.44 (0.77) | 0.45 (0.77)
  SIPD(24) | 12.06 (3.01) | 5.80 (3.00) | 13.08 (3.03) | 24.65 (3.68) | 2.26 (3.67)
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; SPID(6): LS mean estimate of the treatment difference along with 90% confidence interval (CI) were based on an ANCOVA model included treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS Mean Difference = 2.07, 90% CI 2-sided [0.43 to 3.71], Standard Error of Mean 0.99
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; SPID(6): LS mean estimate of the treatment difference along with 90% CI were based on an ANCOVA model included treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS Mean Difference = 1.69, 90% CI 2-sided [0.05 to 3.33], Standard Error of Mean 0.99
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 2.34, 90% CI 2-sided [0.69 to 3.99], Standard Error of Mean 1.00
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; LS Mean Difference = 6.99, 90% CI 2-sided [5.19 to 8.79], Standard Error of Mean 1.09
Statistical Analysis 5: Comparison: PF-05089771 150 mg vs Placebo; SPID(24): LS mean estimate of the treatment difference along with 90% CI were based on an ANCOVA model included treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS Mean Difference = 9.80, 90% CI 2-sided [1.97 to 17.63], Standard Error of Mean 4.74
Statistical Analysis 6: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 3.55, 90% CI 2-sided [-4.28 to 11.37], Standard Error of Mean 4.74
Statistical Analysis 7: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 10.82, 90% CI 2-sided [2.97 to 18.68], Standard Error of Mean 4.76
Statistical Analysis 8: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; LS Mean Difference = 22.39, 90% CI 2-sided [13.82 to 30.97], Standard Error of Mean 5.19

6. Secondary Outcome: Total Pain Relief From 0 to 24 Hours (TOTPAR[24])
Description: TOTPAR(24) was defined as the total area under the PR curve through the first 24 hours after dosing, calculated using trapezoidal rule. PR was assumed to be 0 at 0 hour. PR assessed on a 5-point categorical scale: 0 (none), 1 (a little), 2 (some), 3 (a lot) and 4 (complete), at different time points during the study up to 6 hours. Total score range for TOTPAR (24): 0 (worst) to 96 (best), higher value indicated greater degree of PR. The least square mean and standard error are based on ANCOVA model with treatment as a fixed effect and baseline pain intensity as a covariate
Time Frame: 0 to 24 hours
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
units on a scale | 30.89 (4.23) | 22.81 (4.22) | 31.19 (4.26) | 51.18 (5.17) | 18.63 (5.16)
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; LS mean estimate of the treatment difference along with 90% CI were based on an ANCOVA model including treatment as a fixed effect and baseline pain intensity as a covariate; Test type: Superiority or Other; LS Mean Difference = 12.26, 90% CI 2-sided [1.26 to 23.27], Standard Error of Mean 6.66
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; LS Mean Difference = 4.18, 90% CI 2-sided [-6.82 to 15.18], Standard Error of Mean 6.66
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; Test type: Superiority or Other; LS Mean Difference = 12.57, 90% CI 2-sided [1.52 to 23.61], Standard Error of Mean 6.69
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; Test type: Superiority or Other; LS Mean Difference = 32.56, 90% CI 2-sided [20.51 to 44.61], Standard Error of Mean 7.30

7. Secondary Outcome: Time to Onset of First Perceptible Pain Relief
Description: Participants evaluated the time to first perceptible pain relief by stopping a stopwatch labeled 'first perceptible pain relief' at the moment they first began to experience any relief.
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
hours | 0.6 [0.3 to 0.8] | 0.3 [0.3 to 0.5] | 0.4 [0.3 to 0.7] | 0.5 [0.3 to 0.6] | 0.7 [0.3 to 1.0]
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; Hazard Ratio (HR) estimates of the treatment difference along with 90% CI were based on Cox proportional hazards model including treatment and baseline pain intensity as fixed effects; Test type: Superiority or Other; Hazard Ratio (HR) = 1.0, 90% CI 2-sided [0.6 to 1.5]
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; HR estimates of the treatment difference along with 90% CI were based on Cox proportional hazards model including treatment and baseline pain intensity as fixed effects; Test type: Superiority or Other; Hazard Ratio (HR) = 1.3, 90% CI 2-sided [0.9 to 1.9]
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.1, 90% CI 2-sided [0.7 to 1.6]
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.6, 90% CI 2-sided [1.0 to 2.4]

8. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Participants evaluated the time to first meaningful relief by stopping a stopwatch labeled 'meaningful pain relief' at the moment they first began to experience meaningful relief.
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
hours | 3.3 [2.5 to 4.0] | 2.7 [2.1 to 3.2] | 3.7 [2.6 to 4.7] | 1.3 [0.8 to 1.8] | 4.6 [2.9 to NA] — The upper limit of 90% CI was not calculable because of censored data.
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 2.0, 90% CI 2-sided [1.1 to 3.8]
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 2.6, 90% CI 2-sided [1.4 to 4.9]
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 2.2, 90% CI 2-sided [1.1 to 4.1]
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 5.3, 90% CI 2-sided [2.8 to 9.9]

9. Secondary Outcome: Time to First Use of Rescue Medication
Description: Time to first use of rescue medication (acetaminophen 500 mg or hydrocodone 5 mg) was calculated by subtracting time of first administration of study medication from the rescue medication administration time.
Time Frame: 0 to 24 hours
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
hours | 4.0 [2.4 to 6.6] | 2.5 [2.3 to 3.7] | 5.5 [2.5 to 10.1] | 12.1 [8.9 to NA] — The upper limit of 90% CI was not calculable because of censored data. | 2.3 [1.8 to 2.6]
Statistical Analysis 1: Comparison: PF-05089771 150 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.6, 90% CI 2-sided [0.4 to 1.0]
Statistical Analysis 2: Comparison: PF-05089771 450 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 90% CI 2-sided [0.5 to 1.2]
Statistical Analysis 3: Comparison: PF-05089771 1600 mg vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.5, 90% CI 2-sided [0.3 to 0.8]
Statistical Analysis 4: Comparison: Ibuprofen vs Placebo; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.4, 90% CI 2-sided [0.2 to 0.6]

10. Secondary Outcome: Number of Participants With Global Evaluation of Study Medication
Description: Participant rated the study medication at 6 hours, 24 hours and immediately prior to rescue medication intake (only for participants who took rescue medication[RM]), on 5-point categorical scale: 1=poor, 2=fair, 3=good, 4=very good, and 5=excellent.
Time Frame: 6, 24 hours, prior to rescue medication (assessed up to 24 hours)
Population: FAS: all randomized participants who received >=1 dose of study treatment, had >=1 evaluable (>=90 minutes post-dose) PR score. Participants who received RM prior to 90 minutes were not included in FAS. N(number of participants analyzed): participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
participants
  Hour 6: Poor: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  Hour 6: Poor | 2 | 0 | 3 | 2 | 0
  Hour 6: Fair: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  Hour 6: Fair | 6 | 3 | 3 | 1 | 2
  Hour 6: Good: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  Hour 6: Good | 11 | 9 | 5 | 1 | 5
  Hour 6: Very Good: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  Hour 6: Very Good | 4 | 6 | 11 | 18 | 1
  Hour 6: Excellent: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  Hour 6: Excellent | 2 | 2 | 3 | 7 | 0
  Hour 24: Poor: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  Hour 24: Poor | 0 | 0 | 2 | 0 | 0
  Hour 24: Fair: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  Hour 24: Fair | 2 | 1 | 2 | 0 | 0
  Hour 24: Good: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  Hour 24: Good | 7 | 5 | 2 | 1 | 4
  Hour 24: Very Good: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  Hour 24: Very Good | 5 | 5 | 5 | 7 | 3
  Hour 24: Excellent: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  Hour 24: Excellent | 3 | 1 | 9 | 6 | 0
  Prior to RM: Poor: number analyzed (Participants) | 37 | 42 | 34 | 22 | 29
  Prior to RM: Poor | 26 | 26 | 21 | 6 | 22
  Prior to RM: Fair: number analyzed (Participants) | 37 | 42 | 34 | 22 | 29
  Prior to RM: Fair | 7 | 7 | 9 | 1 | 6
  Prior to RM: Good: number analyzed (Participants) | 37 | 42 | 34 | 22 | 29
  Prior to RM: Good | 4 | 5 | 3 | 3 | 1
  Prior to RM: Very Good: number analyzed (Participants) | 37 | 42 | 34 | 22 | 29
  Prior to RM: Very Good | 0 | 3 | 1 | 6 | 0
  Prior to RM: Excellent: number analyzed (Participants) | 37 | 42 | 34 | 22 | 29
  Prior to RM: Excellent | 0 | 1 | 0 | 6 | 0

11. Secondary Outcome: Number of Participants With Study Medication Satisfaction
Description: Participants provided assessment regarding satisfaction with study medication (SM) for pain relief (PR) and overall performance (OP) on a 5-point categorical scale, 1=very dissatisfied (VD), 2=somewhat dissatisfied (SD), 3=neither satisfied nor dissatisfied (NSND), 4=somewhat satisfied (SS) and 5=very satisfied (VS).
Time Frame: 6, 24 hours, prior to rescue medication (assessed up to 24 hours)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 54 | 54 | 53 | 36 | 36
participants
  SM OP, Hour 6: VS: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM OP, Hour 6: VS | 5 | 6 | 12 | 17 | 0
  SM OP, Hour 6: SS: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM OP, Hour 6: SS | 11 | 9 | 7 | 9 | 6
  SM OP, Hour 6: NSND: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM OP, Hour 6: NSND | 4 | 4 | 2 | 1 | 1
  SM OP, Hour 6: SD: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM OP, Hour 6: SD | 3 | 1 | 2 | 2 | 1
  SM OP, Hour 6: VD: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM OP, Hour 6: VD | 2 | 0 | 2 | 0 | 0
  SM OP, Hour 24: VS: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM OP, Hour 24: VS | 7 | 5 | 13 | 7 | 1
  SM OP, Hour 24: SS: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM OP, Hour 24: SS | 6 | 4 | 3 | 6 | 5
  SM OP, Hour 24: NSND: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM OP, Hour 24: NSND | 3 | 3 | 1 | 0 | 1
  SM OP, Hour 24: SD: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM OP, Hour 24: SD | 1 | 0 | 1 | 0 | 0
  SM OP, Hour 24: VD: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM OP, Hour 24: VD | 0 | 0 | 2 | 1 | 0
  SM OP, Prior to RM: VS: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM OP, Prior to RM: VS | 0 | 4 | 1 | 8 | 0
  SM OP, Prior to RM: SS: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM OP, Prior to RM: SS | 4 | 3 | 3 | 5 | 0
  SM OP, Prior to RM: NSND: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM OP, Prior to RM: NSND | 9 | 5 | 3 | 2 | 4
  SM OP, Prior to RM: SD: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM OP, Prior to RM: SD | 7 | 8 | 7 | 3 | 8
  SM OP, Prior to RM: VD: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM OP, Prior to RM: VD | 16 | 22 | 20 | 4 | 17
  SM PR, Hour 6: VS: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM PR, Hour 6: VS | 5 | 5 | 12 | 18 | 0
  SM PR, Hour 6: SS: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM PR, Hour 6: SS | 9 | 11 | 7 | 9 | 6
  SM PR, Hour 6: NSND: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM PR, Hour 6: NSND | 4 | 1 | 1 | 0 | 0
  SM PR, Hour 6: SD: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM PR, Hour 6: SD | 5 | 3 | 3 | 2 | 2
  SM PR, Hour 6: VD: number analyzed (Participants) | 25 | 20 | 25 | 29 | 8
  SM PR, Hour 6: VD | 2 | 0 | 2 | 0 | 0
  SM PR, Hour 24: VS: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM PR, Hour 24: VS | 7 | 4 | 13 | 10 | 0
  SM PR, Hour 24: SS: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM PR, Hour 24: SS | 4 | 6 | 3 | 3 | 6
  SM PR, Hour 24: NSND: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM PR, Hour 24: NSND | 4 | 2 | 0 | 0 | 1
  SM PR, Hour 24: SD: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM PR, Hour 24: SD | 2 | 0 | 2 | 0 | 0
  SM PR, Hour 24: VD: number analyzed (Participants) | 17 | 12 | 20 | 14 | 7
  SM PR, Hour 24: VD | 0 | 0 | 2 | 1 | 0
  SM PR, Prior to RM: VS: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM PR, Prior to RM: VS | 0 | 3 | 1 | 9 | 0
  SM PR, Prior to RM: SS: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM PR, Prior to RM: SS | 5 | 5 | 1 | 3 | 0
  SM PR, Prior to RM: NSND: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM PR, Prior to RM: NSND | 3 | 4 | 3 | 3 | 3
  SM PR, Prior to RM: SD: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM PR, Prior to RM: SD | 7 | 7 | 9 | 4 | 9
  SM PR, Prior to RM: VD: number analyzed (Participants) | 36 | 42 | 34 | 22 | 29
  SM PR, Prior to RM: VD | 21 | 23 | 20 | 3 | 17

12. Secondary Outcome: Plasma PF-05089771 Concentration
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 10, 24 hours post-dose
Population: Pharmacokinetic analysis set included all randomized participants who received study treatment and had a pharmacokinetic sample analyzed within the treatment period.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg
Number analyzed (Participants) | 55 | 54 | 54
nanogram per milliliter (ng/mL)
  0 hour | NA (NA) — Data was not reported since none of the participants had plasma concentration values above lower limit of quantification (LLOQ). | NA (NA) — Data was not reported since none of the participants had plasma concentration values above lower limit of quantification (LLOQ). | NA (NA) — Data was not reported since none of the participants had plasma concentration values above lower limit of quantification (LLOQ).
  0.5 hour | 1383 (1148.6) | 3497 (3111.2) | 6718 (5774.4)
  1 hour | 3283 (2614.7) | 7770 (5928.5) | 17890 (13217)
  2 hours | 5647 (4144.6) | 14470 (10612) | 31260 (17354)
  4 hours | 4831 (2436.8) | 14110 (7966.7) | 33760 (18706)
  6 hours | 3826 (2261.7) | 11410 (6389.5) | 31390 (16894)
  8 hours | 2874 (1574.3) | 9818 (5280.2) | 29830 (16355)
  10 hours | 2007 (1195.5) | 7916 (4018.3) | 24010 (13993)
  24 hours | 498.0 (344.82) | 2115 (1394.6) | 8521 (5388.1)

13. Secondary Outcome: Plasma Ibuprofen Concentration
Description: Ibuprofen concentration was reported separately for 2 isomers of ibuprofen: (S)-Ibuprofen, and (R)-Ibuprofen, where S implied sinister (clockwise configuration) and R implied rectus (anti-clockwise configuration).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 10, 24 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Ibuprofen
Number analyzed (Participants) | 36
microgram per milliliter (mcg/mL)
  (R)-Ibuprofen 0 hour | 0.0054 (0.0325)
  (R)-Ibuprofen 0.5 hour | 5.510 (6.3603)
  (R)-Ibuprofen 1 hour | 7.049 (6.8608)
  (R)-Ibuprofen 2 hours | 9.042 (6.3054)
  (R)-Ibuprofen 4 hours | 6.522 (4.7188)
  (R)-Ibuprofen 6 hours | 2.574 (2.3774)
  (R)-Ibuprofen 8 hours | 1.081 (1.4523)
  (R)-Ibuprofen 10 hours | 0.4424 (0.5976)
  (R)-Ibuprofen 24 hours | 0.0768 (0.4028)
  (S)-Ibuprofen 0 hour | NA (NA) — Data was not reported since none of the participants had plasma concentration values above lower limit of quantification (LLOQ).
  (S)-Ibuprofen 0.5 hour | 4.343 (5.0224)
  (S)-Ibuprofen 1 hour | 5.623 (5.4780)
  (S)-Ibuprofen 2 hours | 7.356 (4.9376)
  (S)-Ibuprofen 4 hours | 9.638 (4.1646)
  (S)-Ibuprofen 6 hours | 6.039 (3.1734)
  (S)-Ibuprofen 8 hours | 3.597 (2.4122)
  (S)-Ibuprofen 10 hours | 1.955 (1.6135)
  (S)-Ibuprofen 24 hours | 0.1041 (0.4332)

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to 28 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Day 28 (follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 55 | 54 | 54 | 36 | 36
participants
  Adverse Events | 22 | 24 | 28 | 12 | 16
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Findings
Description: Hematology (hemoglobin, hematocrit, red blood cell count, platelets, leukocytes, total neutrophils, eosinophils, basophils, lymphocytes, monocytes), blood chemistry (total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, creatinine, blood urea nitrogen, fasting glucose, uric acid, sodium, potassium, chloride, bicarbonate, calcium, albumin, total protein, creatine kinase), and urinalysis (urine white blood cells, urine red blood cells) were performed.
Time Frame: Baseline up to Day 7 to 10 (follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 55 | 54 | 54 | 36 | 36
participants | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Clinically significant vital signs: supine/sitting pulse rate (PR) less than (<) 40 or more than (>) 120 beats per minute (bpm), standing PR <40 or >140 bpm; systolic blood pressure (BP) >=30 millimeters of mercury (mmHg) change from baseline; absolute systolic BP <90 mmHg; diastolic BP >=20 mmHg change from baseline; absolute systolic BP <50 mmHg.
Time Frame: Baseline up to Day 7 to 10 (follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 55 | 54 | 54 | 36 | 36
participants | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Clinically significant ECG abnormalities: PR interval >=300 milliseconds (msec); 25% increase from baseline in PR interval when baseline PR was >200 msec; an increase from baseline of >=50% in PR interval when baseline PR was <=200 msec; QRS interval >=140 msec; an increase from baseline of >=50% in QRS interval; corrected QT interval (QTc) >=500 msec.
Time Frame: Baseline up to Day 7 to 10 (follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Number analyzed (Participants) | 55 | 54 | 54 | 36 | 36
participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-05089771 150 mg | PF-05089771 450 mg | PF-05089771 1600 mg | Ibuprofen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/54 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 16/55 | 20/54 | 23/54 | 10/36 | 12/36
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05089771 150 mg (N=55) | PF-05089771 450 mg (N=54) | PF-05089771 1600 mg (N=54) | Ibuprofen (N=36) | Placebo (N=36)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 11 | 14 | 4 | 4
Vomiting (Gastrointestinal disorders) | 3 | 5 | 9 | 0 | 1
Feeling hot (General disorders) | 1 | 1 | 2 | 0 | 1
Alveolar osteitis (Infections and infestations) | 3 | 2 | 2 | 1 | 3
Tooth infection (Infections and infestations) | 0 | 0 | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 7 | 8 | 2 | 2
Headache (Nervous system disorders) | 8 | 3 | 5 | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.